CLINICAL TRIAL: NCT02358083
Title: Attitudes Toward Human Papillomavirus and Influenza Vaccination Among Mothers of Early Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Gregory Zimet, Professor, Indiana University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 8645194
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Human Papillomavirus Vaccines; Influenza Vaccines; Attitude to Health
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (12):
- Arm 1. HPV + Control + Control (No Intervention): HPV is target vaccine. No message regarding relative safety of vaccine; Provider provides brief routine recommendation for vaccination.
- Arm 2. HPV + Control + Strong (Experimental): HPV is target vaccine; No message regarding relative safety of vaccine; Provider provides strong recommendation for vaccination.
  Interventions: Behavioral: Provider Communication about Vaccination
- Arm 3. HPV + Control + Disclosure (Experimental): HPV is target vaccine; No message regarding relative safety of vaccine; Provider provides strong recommendation for vaccination and personal disclosure regarding own child's vaccination history.
  Interventions: Behavioral: Provider Communication about Vaccination
- Arm 4. HPV + Safety + Control (Experimental): HPV is target vaccine; Provider provides message about relative safety of vaccination compared to other common daily activities; Provider provides brief routine recommendation for vaccination.
  Interventions: Behavioral: Provider Communication about Vaccination
- Arm 5. HPV + Safety + Strong (Experimental): HPV is target vaccine; Provider provides message about relative safety of vaccination compared to other common daily activities; Provider provides strong recommendation for vaccination.
  Interventions: Behavioral: Provider Communication about Vaccination
- Arm 6. HPV + Safety + Disclosure (Experimental): HPV is target vaccine; Provider provides message about relative safety of vaccination compared to other common daily activities; Provider provides strong recommendation for vaccination and personal disclosure regarding own child's vaccination history.
  Interventions: Behavioral: Provider Communication about Vaccination
- Arm 7. Flu + Control + Control (No Intervention): Flu is target vaccine. No message regarding relative safety of vaccine; Provider provides brief routine recommendation for vaccination.
- Arm 8. Flu + Control + Strong (Experimental): Flu is target vaccine; No message regarding relative safety of vaccine; Provider provides strong recommendation for vaccination.
  Interventions: Behavioral: Provider Communication about Vaccination
- Arm 9. Flu + Control + Disclosure (Experimental): Flu is target vaccine; No message regarding relative safety of vaccine; Provider provides strong recommendation for vaccination and personal disclosure regarding own child's vaccination history.
  Interventions: Behavioral: Provider Communication about Vaccination
- Arm 10. Flu + Safety + Control (Experimental): Flu is target vaccine; Provider provides message about relative safety of vaccination compared to other common daily activities; Provider provides brief routine recommendation for vaccination.
  Interventions: Behavioral: Provider Communication about Vaccination
- Arm 11. Flu + Safety + Strong (Experimental): Flu is target vaccine; Provider provides message about relative safety of vaccination compared to other common daily activities; Provider provides strong recommendation for vaccination.
  Interventions: Behavioral: Provider Communication about Vaccination
- Arm 12. Flu + Safety + Disclosure (Experimental): Flu is target vaccine; Provider provides message about relative safety of vaccination compared to other common daily activities; Provider provides strong recommendation for vaccination and personal disclosure regarding own child's vaccination history.
  Interventions: Behavioral: Provider Communication about Vaccination

INTERVENTIONS:
Behavioral: Provider Communication about Vaccination — There are 12 pairs of messages varying in target vaccination, discussion of relative safety of vaccination, and strength of provider recommendation for vaccination.
  Arms: Arm 10. Flu + Safety + Control; Arm 11. Flu + Safety + Strong; Arm 12. Flu + Safety + Disclosure; Arm 2. HPV + Control + Strong; Arm 3. HPV + Control + Disclosure; Arm 4. HPV + Safety + Control; Arm 5. HPV + Safety + Strong; Arm 6. HPV + Safety + Disclosure; Arm 8. Flu + Control + Strong; Arm 9. Flu + Control + Disclosure

SUMMARY:
The purpose of this study was to determine whether messages about 1. relative risk of vaccination vs. other activities and 2. strength of doctor's recommendation influenced parental intention to get own child vaccinated against human papillomavirus (HPV) or Influenza.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Lives in United States
* Mother or female legal guardian of at least one child aged 9-13
* Able to understand English
* For HPV condition: Target child must not have received any doses of HPV vaccine
* For Flu condition: Target child must not have received the flu vaccine during the prior flu season

Exclusion Criteria:

* Under 18 years of age
* Not mother or female legal guardian of at least one child ages 9-13
* Not living in United States
* Not able to understand English and Spanish
* For HPV condition: Target child had already received at least 1 dose of the HPV vaccine
* For Flu condition: Target child received the influenza vaccine during the previous flu season

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1165 (Actual)
Dates: Start 2014-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Willingness to vaccinate child with target vaccine | During survey administration, at approximately 15 minutes into the survey.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Zimet, PhD, Principal Investigator — Indiana University